CLINICAL TRIAL: NCT06057077
Title: A Randomized Clinical Trial Comparing Semaglutide GLP1 Agonists With Degludec Basal-bolus Insulin in Early Type 1 Diabetes
Brief Title: Semaglutide GLP1 Agonists With Degludec Basal-bolus Insulin in Early Type 1 Diabetes to Basal-bolus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, public health department, MSc, Riaydh first health cluster, Ministry of health , Saudia arabia, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amr Ahmed, Maher M.Akl
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: To compare the efficacy and safety of basal-bolus insulin degludec and semaglutide with the regular standard of care versus basal-bolus insulin with regular standard of care in early type 1 diabetic patients.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 60 early type 1 diabetes with semaglutide and degludec basal bolus insulin (Active Comparator): degludec administered once daily bolus insulin three times daily and time in range and Semaglutide once weekly
  Interventions: Drug: Semaglutide weekly injection
- 60 early type 1 diabetes with degludec basal bolus insulin with regular standard of care (No Intervention): 60 patients' Basal insulin degludec administered once daily according to the SMBG and continuous plan at the clinic bolus insulin three times daily according to the meals and time in range and carbohydrate index Dosing adjusted based on SMBG results

INTERVENTIONS:
Drug: Semaglutide weekly injection — semaglutide is Glp1 AGONIST WHICH IS NEW CHALLENGE IN DIABETES DISEASE TREATMENT EITHER TYPE 2 AND IS APPROVED BY FDA FOE children aged above 12 years at obesity
  Other Names: tresiba once daily
  Arms: 60 early type 1 diabetes with semaglutide and degludec basal bolus insulin

SUMMARY:
type 1 diabetes is an autoimmune disease and still, some unknown mechanisms are undiscovered millions of children and adults suffer from this type which need basal-bolus insulin as the classical regimen, and basal-bolus insulin is the best type of treatment is similar to the physiological pattern, so our target and may studies before how to preserve the residual beta cells or postpone the complete destruction or extend the honeymoon stage to improve quality of life, the most challenge at type 1 diabetes is diabetic ketoacidosis which affect the quality of life and risk of death so at our clinical trials using the combination of basal insulin-like degludec as its action extend to 72 hours and has high flexibility and less hypoglycemic events and has an affinity to 99% to albumin so may be considered the most type of insulin is similar to human physiological insulin as 50% of insulin pass through portal circulation so no insulin until now it is mimic the normal physiological insulin but IDeg is the nearest to normal until now, Objective: To compare the efficacy and safety of basal-bolus insulin degludec and semaglutide with regular standard of care versus basal-bolus insulin with regular standard of care in early type 1 diabetic patients.

In our study, the investigators will compare 2 groups of early type 1 patients in the age group 18 years to 35 years Protocol and Methodology for a Randomized Controlled Trial of Basal-Bolus Insulin Degludec and Semaglutide with Regular Standard of Care Versus Basal-Bolus Insulin with Regular Standard of Care in Early Type 1 Diabetic Patients

Study Design: Randomized, controlled, open-label trial

Setting: Outpatient diabetes clinics

Participants: Early type 1 diabetic patients (aged 18-35 years) who have been diagnosed with type 1 diabetes for less than 2 years and have a hemoglobin A1c (HbA1c) of 7.0-11%.

the tests will be done pre- and post :

1. Anti GAD 65 and anti IA2
2. HA1C
3. Serum C peptide
4. fasting insulin
5. serum zinc

DETAILED DESCRIPTION:
type 1 diabetes is an autoimmune disease and still, some unknown mechanisms are undiscovered millions of children and adults suffer from this type which need basal-bolus insulin as the classical regimen, and basal-bolus insulin is the best type of treatment is similar to the physiological pattern, so our target and may studies before how to preserve the residual beta cells or postpone the complete destruction or extend the honeymoon stage to improve quality of life, the most challenge at type 1 diabetes is diabetic ketoacidosis which affect the quality of life and risk of death so at our clinical trials using the combination of basal insulin-like degludec as its action extend to 72 hours and has high flexibility and less hypoglycemic events and has an affinity to 99% to albumin so may be considered the most type of insulin is similar to human physiological insulin as 50% of insulin pass through portal circulation one of the amazing advantages of IDeg is that no accumulation After 2-3 days of once-daily dosing, IDeg concentrations reach a steady state with no additional accumulation since, at that time, the daily-injected dose equals the daily-eliminated quantity of insulin when repeated equivalent doses are delivered at sufficient intervals.

the tests will be done pre- and post :

1. Anti GAD 65 and anti IA2
2. HA1C
3. Serum C peptide
4. fasting insulin
5. serum zinc

Insulin-bound insulin :

one other advantage of IDeg is insulin-bound insulin so no difference in clearance at renal or liver-impaired patients and normal functions. Albumin-bound insulins are not as easily filtered by the kidney as unbound insulins. Thus, hepatic and renal impairment have no effect on the PK characteristics of these insulin mimics.

synergism between semaglutide as GLP1 agonist and ultralong acting insulin like IDeg is suspected to give more benefits to early type 1 diabetes like extending the honeymoon phase and may preserve the residual beta cells function also may affect autoantibodies like anti-GAD65 and anti islets cells 2 anri IA2 In our study, the investigators will compare 2 groups of early type 1 patients in the age group 18 years to 35 years Protocol and Methodology for a Randomized Controlled Trial of Basal-Bolus Insulin Degludec and Semaglutide with Regular Standard of Care Versus Basal-Bolus Insulin with Regular Standard of Care in Early Type 1 Diabetic Patients

Objective: To compare the efficacy and safety of basal-bolus insulin degludec and semaglutide with regular standard of care versus basal-bolus insulin with regular standard of care in early type 1 diabetic patients.

Study Design: Randomized, controlled, open-label trial

Setting: Outpatient diabetes clinics

Participants: Early type 1 diabetic patients (aged 18-35 years) who have been diagnosed with type 1 diabetes for less than 2 years and have a hemoglobin A1c (HbA1c) of 7.0-11%.

Exclusion Criteria:

Pregnancy or breastfeeding History of severe hypoglycemia History of diabetic ketoacidosis History of pancreatitis History of hypersensitivity to insulin degludec or semaglutide Use of any other antidiabetic medications, other than basal-bolus insulin

Interventions:

Arm 1: Basal-bolus insulin degludec and semaglutide with regular standard of care Arm 2: Basal-bolus insulin with the regular standard of care

Regular standard of care:

Diabetes self-management education Nutritional counseling Physical activity counseling Self-monitoring of blood glucose (SMBG) Insulin dose adjustment Basal-bolus insulin degludec: Administered once daily Dosing adjusted based on SMBG results Semaglutide: Administered once weekly dosing adjusted based on SMBG results

Outcomes:

Primary outcome: Change in HbA1c from baseline to 24 weeks

Secondary outcomes:

Change in body weight from baseline to 24 weeks Frequency of hypoglycemia episodes from baseline to 24 weeks Time in range (TIR) from baseline to 24 weeks Quality of life from baseline to 24 weeks

Sample Size:

A sample size of 120 participants (60 per arm) is estimated to be sufficient to detect a difference of 0.5% in HbA1c between the two arms with a power of 80% and a significance level of 0.05.

Randomization:

Participants will be randomized to one of the two arms using a computer-generated random number table.

Blinding:

The study is open-label, meaning that participants and investigators will be aware of which treatment arm they are in.

Follow-up:

Participants will be followed for 24 weeks. They will be required to attend clinic visits every 6 weeks for assessments of HbA1c, body weight, and frequency of hypoglycemia episodes. They will also be required to wear a continuous glucose monitor (CGM) for 1 week at baseline and at 24 weeks to assess TIR.

Data Analysis:

Data will be analyzed using SPSS software. The primary outcome will be analyzed using an unpaired t-test. Secondary outcomes will be analyzed using appropriate statistical tests, such as chi-squared tests and ANOVA.

Safety:

All participants will be monitored closely for any adverse events. Any adverse events will be reported to the study's safety monitoring committee.

Ethical Considerations:

The study will be conducted in accordance with the Declaration of Helsinki and the International Conference on Harmonization Good Clinical Practice Guidelines. The study protocol will be reviewed and approved by an institutional review board.

Informed Consent:

All participants will be required to provide written informed consent before participating in the study.

Discussion:

This randomized controlled trial will compare the efficacy and safety of basal-bolus insulin degludec and semaglutide with the regular standard of care versus basal-bolus insulin with the regular standard of care in early type 1 diabetic patients. The results of this study will provide valuable information about the best treatment options for this population.

ELIGIBILITY:
Inclusion Criteria:

early diagnosed type 1 diabetic patients were diagnosed in the last 6 months age of two groups: from 18-35 years basal-bolus insulin patients

Exclusion Criteria:

no oral hypoglycemic drugs no pregnancy no hypoglycemic drugs or immunosuppressant no history of diabetic ketoacidosis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
change in HA1c and mounts of insulin of basal and bolus which will be taken daily is the same or decreased after one year of follow up | Time Frame: one year
  change in A1C and daily insulin requirements will be reduced at the end of one year from study was started

SECONDARY OUTCOMES:
the change in weight after follow up of one year | one year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ang JE, Pandher R, Ang JC, Asad YJ, Henley AT, Valenti M, Box G, de Haven Brandon A, Baird RD, Friedman L, Derynck M, Vanhaesebroeck B, Eccles SA, Kaye SB, Workman P, de Bono JS, Raynaud FI. Plasma Metabolomic Changes following PI3K Inhibition as Pharmacodynamic Biomarkers: Preclinical Discovery to Phase I Trial Evaluation. Mol Cancer Ther. 2016 Jun;15(6):1412-24. doi: 10.1158/1535-7163.MCT-15-0815. Epub 2016 Apr 5. PMID 27048952
- [Derived] Ahmed A, Monir Akl M. Exploring a Synergistic Approach: Dual GLP-1 Agonist Combined with Degludec Basal Insulin for Early Type 1 Diabetes Treatment and its Impact on Albumin-Insulin Producing Cells Expression. Adv Pharm Bull. 2024 Jul;14(2):262-265. doi: 10.34172/apb.2024.040. Epub 2024 Mar 18. PMID 39206389